CLINICAL TRIAL: NCT06563492
Title: The Effect of Insoles on Muscle Activation and Gait Parameters in Plantar Fasciitis
Brief Title: The Effect of Insoles in Plantar Fasciitis
Acronym: Insoles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hande YAZICI, Lecturer, Medipol University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: HYAZICI
Record Dates: First submitted 2024-08-19; First posted 2024-08-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; insole; EVA; 3D printer; muscle activation
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVA INSOLES (Active Comparator)
  Interventions: Device: insole
- 3D INSOLES (Active Comparator)
  Interventions: Device: insole

INTERVENTIONS:
Device: insole — evaluation of individuals using different insoles

SUMMARY:
It aims to investigate the effect of two personalized insoles made of different materials designed to reduce pain in individuals with plantar fasciitis on muscle activation and gait parameters at 3-month follow-up.

DETAILED DESCRIPTION:
Plantar Fasciitis (PF) occurs after inflammation and thickening of the fascia, which originates from the medial tuberosity of the calcaneus and runs in the medial plantar part of the foot and has a thick fibrous band structure. It aims to investigate the effect of two personalized insoles made of different materials designed to reduce pain in individuals with plantar fasciitis on muscle activation and gait parameters at 3-month follow-up. The participants of the study will consist of male and female individuals between the ages of 18-65 who are diagnosed with plantar fasciitis by a specialist doctor, who apply to the Prosthetic Orthotics Center (POMER) with a personalized insoles prescription, and who volunteer to participate in the study.Participants will be provided with demographic information, foot function assessment, pedobarographic analysis, gait assessment, muscle activity assessment, and satisfaction assessment. The Foot Function Index (FFI) will be used to assess foot function in individuals with plantar fasciitis. Foot plantar pressure distribution analysis will be performed using the Tekscan software of the EsCoSCAN® pedobarographic assessment device. The plantar pressure analysis and physical evaluation of the individual will be performed and produced by Computer Aided Design and Computer Aided Manufacturing (CAD-CAM) method. Muscle activation data will be recorded with BIOSIGNALSPLUX Researcher Kit brand EMG device. Satisfaction Assessment-Orthotic Prosthesis Users Questionnaire (OPKA-M) will be used. Sensory evaluation will be evaluated with Semmes Weinstein monoflaments. All data will be evaluated by statistical analysis methods.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65,
* Being diagnosed with plantar fasciitis,
* Being prescribed custom insoles,
* Having complaints for at least 3 months,
* Heel pain complaint is at the plantar medial calcaneal tubercle,
* Pain complaint is most evident in the first steps taken in the morning or in the steps after resting,
* Having a Roles and Maudsley score of 3 or 4 in the initial evaluation

Exclusion Criteria:

* Having a body mass index greater than 30 kg/m2,
* Having any cardiopulmonary, dermatological, neurological or orthopedic problems other than plantar fasciitis,
* Having a history of foot or ankle surgery,
* Using an assistive device (walker, canadiens, etc.)
* Not using appropriate shoes,
* Having cognitive, mental and/or psychological problems
* Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2025-01-06 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Electromyography | Change from Baseline of treatment at 3 months
  Muscle activation data will be recorded with BIOSIGNALSPLUX Researcher Kit brand EMG device. EMG is a frequently used method that evaluates muscle activation as a lens. In EMG measurements, signals are classified non-invasively using surface electrodes (20) The electrodes are planned according to the Gluteus Maximus, Gluteus Medius, Rectus Femoris, Biceps Femoris, Gastrocnemius Medialis and Lateralis, Soleus, Tibialis Anterior muscles.

SECONDARY OUTCOMES:
Pedobarographic Analysis | Change from Baseline of treatment at 3 months
  Foot plantar pressure distribution analysis will be performed using the Tekscan software of the EsCoSCAN® pedobarographic evaluation device. In the static analysis; fore-hindfoot loading (kg), total loading (kg), fore-hindfoot weight ratio (%), fore-hindfoot plantar contact surface (cm2), total plantar contact surface (cm2), maximum pressure (kg/cm2), average pressure (kg/cm2), foot center (CoF), foot angle (°) values are obtained. Fore-hindfoot relationship is also evaluated. In dynamic analysis; Fore-hindfoot loading (kg), total loading (kg), foot plantar contact surface (cm2), average pressure (kg/cm2), maximum pressure (kg/cm2), acceleration (cm/s), step length (cm), cadence (step/min) and step width data of the individual are recorded. Fore-hindfoot relationship is also evaluated under dynamic conditions.
Foot Function Index (FFI) | Change from Baseline of treatment at 3 months
  The Foot Function Index (FFI) will be used to assess foot function in individuals with plantar fasciitis. The foot function index is a widely used form that can be completed by the individual and developed to measure the effects of foot pathologies on pain, disability and activity limitation. Yalıman et al. translated and adapted the Foot Function Index to Turkish for patients with plantar fasciitis. It consists of 23 items with 3 subgroups. The pain subscale, which includes 9 items, measures the level of foot pain in various situations, while the disability subscale, which includes 9 items, determines the degree of difficulty in performing various functional activities due to foot problems. The activity limitation subscale, which includes 5 items, evaluates activity limitations due to foot problems.
Satisfaction Evaluation | Change from Baseline of treatment at 3 months
  Orthosis Prosthesis Users Survey (OPKA-M) was developed in 2003. It is used to make quality assessment in the field of orthosis and prosthesis, to maintain awareness of development in activities, to evaluate changes in functional status and quality of life of patients, to evaluate satisfaction with prosthesis orthosis and services. OPKA-M survey is a satisfaction survey developed for upper and lower extremity prosthesis and orthosis users. It consists of 21 questions in total. It is a survey that evaluates satisfaction with the orthosis used and the service received.
Sensory Evaluation | Change from Baseline of treatment at 3 months
  Loss of pressure sensation will be assessed with "Semmes Weinstein" monofilaments. If there is loss of sensation in the assessment made with this filament that applies 10 g pressure to the foot, the patient's foot is at risk and the protective sensation has been lost. The 5.07 nylon monofilament used in the test is manufactured to bend when 10 g force is applied. This pressure is applied to specific points located on the plantar and dorsal sides of the foot.